CLINICAL TRIAL: NCT06912113
Title: The Effect of Motivational Interviewing on Smoking Quit Intention in Lung Cancer Patients: a Randomized Controlled Trial
Brief Title: The Effect of Motivational ınterviewing on ıntention to Quit Smoking in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Sibel Doğru, Assistant professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/92
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Motivational Enhancement; İntention to Quit
Keywords: Motivational enhancement; Real-time video counselling; Lung cancer; İntention to quit smoking
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No intervention was made to this arm, routine maintenance procedure was applied.
- Intervention (Experimental): In this study, an online motivational interview was conducted over the real-time video counselling regarding quitting smoking.
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — What distinguishes this intervention from other clinical applications is that in this study, the clinical effectiveness of motivational interviewing was examined by using a smoking cessation intention scale before and after the intervention.
  Arms: Intervention

SUMMARY:
The effect of online video conferencing on smoking cessation intention in patients diagnosed with lung cancer was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18,
* diagnosed with lung cancer, who had smoked at least 100 cigarettes in their lifetime and had smoked at least one cigarette in the last month,
* who volunteered to participate in the study,
* who had no communication problems, and who had internet access were included in the study.

Exclusion Criteria:

* Occasional smokers,
* Those using a different type of nicotine than cigarettes,
* Those actively participating in other smoking cessation programs, and those reporting dependence on any medication were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Intention to quit smoking scale | Four weeks
  It was developed by Söyler et al. to measure the intention to quit smoking in smokers and consists of eight questions. The scoring of the scale is carried out by summing the scores obtained for each item. The scale includes the following questions: 1. I plan to quit smoking, 2. I will try to quit smoking, 3. I dream about quitting smoking, 4. I want to quit smoking, 5. Quitting smoking is important to me, 6. I will quit smoking soon, 7. I am doing research on quitting smoking, 8. I intend to meet with a health professional about quitting smoking. The questions in the scale were evaluated with a five-point Likert. Cronbach's alpha value is 0.929. The minimum score that can be obtained from the scale is 8, and the maximum score is 40. Increasing scores indicate an increasing intention to quit smoking, while decreasing scores indicate a decreasing intention to quit smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided